CLINICAL TRIAL: NCT03159026
Title: Chart Review of Patients Who Have the Amish/Mennonite Variant of Propionic Acidemia
Brief Title: Review of Charts From Amish/Mennonite Variant PA Patients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Lina Ghaloul Gonzalez, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO16110176
Record Dates: First submitted 2017-04-12; First posted 2017-05-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Propionic Acidemia
Keywords: Amish/Mennonite variant
MeSH Terms: conditions — Propionic Acidemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The natural history of patients with PA-AMV has not been systematically studied before and there is no published data in the literature about this condition since 1980. There is no evidence-based approach to care of these patients, particularly the younger patients who may no come to medical attention until significant cardiac problems develop. Through systematic review of existing medical records on essentially all known patient with this condition, investigators plan to develop an evidence-based management plan for preventive care of these patients.

DETAILED DESCRIPTION:
The study is designed to provide a comprehensive description of the clinical and biochemical features of propionic academia, Amish/Mennonite variant (PA-AMV). From these data, the investigators hope to identify biomarkers for assessment of clinical course and efficacy of ongoing management.

The investigators plan to identify essentially all known patients who have the Amish/Mennonite variant of Propionic academia (PA-AMV) through collaboration with clinicians who proved care to this extended community. Signed consents include permission to access life-long medical records to allow investigators to define the natural history of this biochemical variant condition. This will include a description the clinical and biochemical features and natural history of patients with propionic acidemia in the Amish/Mennonite population. In particular, there is interest in the cardiac complications of this variant, so investigators will analyze EKG, echo and cardiac MRI findings in above patients. These data will be used to Identify biomarkers for clinical assessment and ongoing management.

There has been no published data on patients with PA-AMV since 1980. Accumulated clinical experience with PA Amish/Mennonite variant patients suggests that these patients tend to have less severe clinical features compared to classic PA. Severe neonatal metabolic decompensation and ketoacidosis are not present in Amish/Mennonite patients we have followed. Describing the natural history and clinical course is essential in this group of patients to further guide their management. There is currently no evidence-based approach to care of these patients, but rather individual medical centers manage patients symptomatically and differently. A uniform, data-driven approach to patient management is needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients homozygous for the PCCB c.606A>G mutation

Exclusion Criteria:

* Patients who are not homozygous for the PCCB c.1606A>G mutation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Amish and Mennonite individuals who have been diagnosed as having the PA-AMV form of propionic academia as characterized by the presence of homozygous PCCB c.1060A>G.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Clinical and biochemical natural history of Amish/Mennonite PA variant | Through study completion, an average of one year.
  Chart review to describe clinical and biochemical features of Amish/Mennonite PA variant

CONTACTS AND LOCATIONS:
Overall Officials: Lina Ghaloul-Gonzalez, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No